CLINICAL TRIAL: NCT03175380
Title: Collection and Storage of Biological Samples Obtained by Leukapheresis for the Future Study of Immune Responses Induced by Two BCG Vaccinations in BCG-naïve Healthy Adults in the US (A-051)
Brief Title: Biological Samples Obtained by Leukapheresis Induced by Two BCG Vaccinations in BCG-naïve Healthy Adults in the US
Acronym: (A-051)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A-051
Record Dates: First submitted 2017-04-17; First posted 2017-06-05 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: All participants (N=17) will receive BCG on Study Day 0 and Study Day 180 by intradermal administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bacillus Calmette-Guérin (Experimental): All participants will receive a total of two doses of bacillus Calmette-Guérin (BCG), by intradermal injection, approximately 6 months apart. They will be observed for 284 days
  Interventions: Biological: bacillus Calmette-Guérin

INTERVENTIONS:
Biological: bacillus Calmette-Guérin — BCG injection for prevention of tuberculosis
  Other Names: BCG

SUMMARY:
This protocol will use leukapheresis to collect lymphocytes to study immune responses following vaccination with BCG in BCG-naïve participants. These studies will include, but not necessarily be limited to: anti-T-cell and anti-Natural Killer (NK) T-cell responses, anti-lipid responses, and antibody responses to BCG following re-vaccination. These responses will provide a detailed framework characterizing the immune responses that are induced and responses that are not induced in humans by BCG, a partially protective TB vaccine. This framework will allow new hypotheses to be formulated and tested regarding what new and more effective TB vaccines should target for optimal protective immunity.

DETAILED DESCRIPTION:
This is an open-label protocol in up to 15 healthy adults who are BCG-naïve. All participants will receive a total of two doses of BCG, by intradermal injection, approximately 6 months apart. Participants will be followed by a combination of visits and telephone contacts through Study Day 264. Participants will undergo TST testing 3 months after the second BCG vaccination and QuantiFERON TB Gold in-Tube (QTBGT), or the equivalent, if necessary. Two BCG vaccinations given 6 months apart were chosen for this study to give optimal T cell and antibody responses for future study. Leukapheresis will be conducted prior to the first BCG vaccination and at 56 days after the second BCG vaccination (Hoft, 2002; Brown, 2003; de Valliere, 2005). The final leukapheresis timing was selected based on results from functional biological assays, which suggest analysis of samples at this time point may provide insight into the protective immune responses elicited by BCG, and on results of prior clinical trials describing the peak immune responses to BCG (Hoft, 2002; Brown, 2003; de Valliere, 2005). The study will be conducted at a single site in the US (Saint Louis University [SLU]).

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent process.
2. Is age ≥18 years and ≤55 years on Study Day 0.
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study.
4. Agrees to avoid elective surgery during the study.
5. Willingness to receive HIV test results.
6. For female participants: agrees to avoid pregnancy from 21 days prior to Study Day 0 and for the full duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide.
7. Has general good health, confirmed by medical history and physical examination.
8. Has not received vaccination or immunotherapy with a BCG product at any time prior to Study Day 0.
9. Body weight of > 110 pounds
10. Absence of previous risk factors for HIV infection including:

    * History of IV drug abuse
    * History of unprotected intercourse with known HIV infected individual
    * Men having sex with men

Exclusion Criteria:

Participants must have none of the following at the time of study entry:

1. Acute illness on Study Day 0.
2. HIV-1/2 positive
3. Oral temperature ≥37.5°C on Study Day 0.
4. Abnormal laboratory values per local laboratory parameters from most recent blood collection prior to Study Day 0 as follows:

   * hemoglobin, hematocrit, absolute neutrophil count, or absolute lymphocyte count below lower limit of normal (LLN)
   * white blood cell count above upper limit of normal (ULN) or below LLN (i.e., must be within normal limits)
   * ALT, AST, GGT, total bilirubin, alkaline phosphatase (ALP), blood urea nitrogen (BUN), creatinine >1.25 times institutional upper limit of normal
   * Calcium not within institutional normal limits
   * Fibrinogen level <100 mg/dL.
5. Evidence of significant active infection.
6. Evidence of central nervous system tuberculosis or pleural tuberculosis.
7. Positive QuantiFERON TB Gold in-Tube (or equivalent).
8. History of treatment for active or latent tuberculosis infection.
9. History or evidence of active tuberculosis.
10. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis.
11. History of occupational exposure to an individual with active tuberculosis in a health care setting.
12. History of autoimmune disease or immunosuppression.
13. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted).
14. Received immunoglobulin or blood products within 42 days before Study Day 0.
15. Received any investigational drug or investigational vaccine within 182 days before Study Day 0, or planned participation in any other interventional study during the study period.
16. Received investigational TB vaccine at any time.
17. Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 56 days after the last BCG vaccination in this study.
18. Current chronic drug therapy including hormone replacement such as thyroxin, insulin, etc. (estrogen and progesterone replacement and contraceptives are acceptable).
19. History or laboratory evidence of any past, present, or future possible immunodeficiency state including but not limited to any laboratory indication of HIV-1 infection.
20. Any contraindications for BCG administration as described in the BCG package insert (Appendix B).
21. Previous medical history that may compromise the safety of the participant in the study, including but not limited to: severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy.
22. Evidence of a new acute illness that may compromise the safety of the participant in the study.
23. History or evidence of chronic hepatitis.
24. History of alcohol or drug abuse within the past 2 years.
25. History of keloid formation.
26. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of BCG, including axillary lymphadenopathy.
27. All female participants: currently pregnant or lactating/nursing; or positive urine pregnancy test during screening, on the day of BCG vaccination.
28. History of being deferred as a blood donor because of problems associated with tolerating the procedure.
29. Having donated > 120 mL of blood within the last 8 weeks.
30. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol.
31. In the opinion of the investigator and the infusion center team, condition of the participant's veins is not suitable for leukapheresis procedure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Biological samples | 8 months
  Obtain biological samples through leukapheresis and cryopreservation of cells for the future study, by in vitro assay, of immune responses after two doses of BCG in BCG-naïve healthy adults.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hoft, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No